CLINICAL TRIAL: NCT00902629
Title: Randomized Clinical Trial Investigating the Longterm Results of Early vs. Delayed Surgery for Epiretinal Fibrosis.
Brief Title: Epiretinal Fibrosis, Effect of Early Surgery
Acronym: epitell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Mads Kofod, Md, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPITELL
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal Fibrosis; Macular Pucker
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group contains the patients randomized for early treatment of their epiretinal fibrosis.
  Interventions: Procedure: Early surgery
- Control (No Intervention): Control contains patients not randomized for early surgery.

INTERVENTIONS:
Procedure: Early surgery — Intervention group contains patients randomized to receive surgery for their epiretinal fibrosis, at an earlier point than what the common clinical practice is now.
  Arms: Intervention

SUMMARY:
The goal of this randomized clinical trial is to investigate when it is optimal to treat the eye disease epiretinal fibrosis.

Hypothesis: In a population of patients with symptomatic idiopathic epiretinal fibrosis and visual acuity above 0.4, the best long term outcome measured by visual acuity is achieved by early surgery compared to periodic controls until a continual loss of visual acuity has been ensure followed by surgery.

DETAILED DESCRIPTION:
Epiretinal fibrosis is a disease of the macula, which affects the central retina, and there by the central vision. Epiretinal fibrosis is due to a growth of connective tissue on retinas surface.

From population studies shows that 15% of patients with epiretinal fibrosis will develop moderate to severe loss of visual acuity. Earlier studies have shown that surgery to remove the epiretinal membrane most often leads to improvements in visual acuity if not a normalization of this. The reason why not everyone has normalization of their visual acuity could be growth of connective in the deeper layers of the retina. This intraretinal fibrosis develops over time and is presumed to worsen with the duration of the condition.

In a patient with symptomatic epiretinal fibrosis and visual acuity over 0,4, the current clinical practice is to utilize the wait and see approach, where you hold of treatment until you have made sure that the patients visual acuity is declining. With the wait and see approach you avoid doing surgery on eyes that would have remained stable in their visual acuity. On the other hand will the same approach always ensure that we do surgery on eye that have deteriorated visual acuity, usually to a point of 0,1-0,3 and longer duration of disease.

Hence the results of delayed surgery are presumably worse than what could have been achieved by operating at an earlier point.

This project aims to investigate if you can give the patients a more favorable long term result by doing surgery earlier compared to the traditional wait and see approach.

This study is a prospective randomized clinical trial. We aim to include 60 patients, where 20 will be randomized to early surgery (intervention) and 40 to a close follow-up program(control). If the patients in the control group loss more than 10 Early Treatment Diabetic Retinopathy Study (ETDRS) letters during the follow-up of of they request surgery for their epiretinal fibrosis they will be offered the same operation as the intervention group.

The Intervention group is to have clear lens extraction if they are not already operated for cataract. This is within 4 weeks of inclusion, and another 4 weeks after this they will have their epiretinal fibrosis removed by pars plana vitrectomy.

There are clinical controls after 3,6,9 and 12 months after inclusion/surgery for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjective loss of visual acuity and/or visual distortions
* Visual acuity more than or equal to 35 ETDRS letters (at 4 meter)
* Duration of symptoms Less than 13 months
* Metamorphopsia on a Amsler Grid
* Binocular vision disturbed

Exclusion Criteria:

* Diabetic eye symptoms
* Previous oculary surgery, except cataract
* Presence of hard drusen in age-related macular degeneration (AMD)
* Other serious eye diseases
* Patients unable to complete the follow up
* not legal guardian of themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in best corrected visual acuity, 12 months after enrollment | 12 months after enrollment

SECONDARY OUTCOMES:
Retinal morphology in the control cohort, 12 months after enrollment | 12 months after enrollement
Change in subjective quality of life 12 month after enrollment. | 12 months after enrollment
Changes in visual field 12 months after enrollment | 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Mads Kofod, MD, Principal Investigator — Eye department, Glostrup University Hospital
Locations (1):
- Eye department, Glostrup University hospital, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Kofod M, Christensen UC, la Cour M. Deferral of surgery for epiretinal membranes: Is it safe? Results of a randomised controlled trial. Br J Ophthalmol. 2016 May;100(5):688-92. doi: 10.1136/bjophthalmol-2015-307301. Epub 2015 Sep 16. PMID 26377411